CLINICAL TRIAL: NCT05624892
Title: The Effect of Mirror Therapy With Virtual Reality Application on Motor-Sense Acquisition and Quality of Live in Home Care of Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Muhammet Ali AYDIN, Research Assistant, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ATAUNI-001
Record Dates: First submitted 2022-10-13; First posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Stroke Syndrome
Keywords: Stroke; Home Care; Mirror Therapy; Virtual Reality; Nursing
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: In the study, 60 individuals, including 1 experimental and 1 control group, were included in the study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Application of mirror therapy to the experimental group with virtual reality application
  Interventions: Diagnostic Test: Mirror Therapy with Virtual Reality Application
- Control Group (No Intervention): Application of classical mirror therapy to the control group

INTERVENTIONS:
Diagnostic Test: Mirror Therapy with Virtual Reality Application — Researchers will apply Mirror Therapy with Virtual Reality Application to increase individuals' quality of life and motor sense gains.
  Arms: Experimental Group

SUMMARY:
: Aim: Stroke is increasing day by day in our country as in the world. Early rehabilitation after stroke accelerates motor-sensory gains of individuals. This also increases the quality of life. Although there are studies on post-stroke rehabilitation in our country, rehabilitation applications with virtual reality application are very limited. For this reason, the research was carried out to determine the effect of home therapy with virtual reality application on motor-sensory gains and quality of life after stroke.

Material and method: The research was conducted as a randomized controlled experimental study. The universe of the research; Between December 2021 and May 2022, individuals who met the criteria for inclusion in the study who applied for home care to Erzurum Atatürk University Health Application and Research Center Physical Therapy Unit with the diagnosis of loss of movement in the upper extremity after stroke were formed. The sample size for the research was determined by power analysis. In the power analysis, it was determined that a total of 52 people should be reached in order to reach the 95% confidence level at the 0.05 significance level and 80% power at the p<0.05 significance level. Considering that there may be data losses in the study, it was decided to reach 60 people, 15% more than the sample. "Descriptive Feature Form", "Brunnstrom Staging" and "SF-36 Quality of Life Scale" were used to collect data.In the analysis of data; percentile distribution, chi-square, Fisher-Freeman- Halton Exact test, t-test in independent groups, Repeated Measures ANOVA Test, Friedman Test, One Way ANOVA test, Kruskall Wallis test, and post hoc analyzes (Bonferroni, Games Howell, Dunn) were used.

ELIGIBILITY:
Inclusion Criteria:

* Being literate,
* Be over 18 years old,
* Having sufficient communication skills to be able to answer verbal and written questions and follow instructions,
* To have applied to benefit from home care services,
* Having been diagnosed with stroke and being at least 6 days old,
* Not having advanced vision problems,
* Not having a vertigo problem
* Not being diagnosed with epilepsy
* In Brunnstrom staging, Upper extremity Stage 2 and above

Exclusion Criteria:

* To reside outside the borders of Erzurum province
* Be under the age of 18
* In Brunnstrom staging, the upper extremity is below Stage 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Rehabilitation of the experimental and control groups for 30 minutes 3 days a week for 4 weeks | One month
  Individuals in the experimental and control groups were evaluated with the "Brunnstrom Staging" and the "SF-36 Quality of Life Scale". The Brunnstrom Staging" and the "SF-36 Quality of Life Scale consists of 8 sub-dimensions. It is expected that the average score will increase in all sub-dimensions of the scale. Higher scores indicate that physical function, social functionality, mental health, energy/vitality and general health sub-dimensions increase. Similarly, higher scores indicate a decrease in physical role difficulty, emotional role difficulty and pain.

SECONDARY OUTCOMES:
Collection of the final test | Three monts
  The final test for individuals in the experimental and control groups were evaluated with the "Brunnstrom Staging" and the "SF-36 Quality of Life Scale". The experimental group received mirror therapy with virtual reality application, and the control group had classical mirror therapy. The Brunnstrom Staging" and the "SF-36 Quality of Life Scale consists of 8 sub-dimensions. It is expected that the average score will increase in all sub-dimensions of the scale. Higher scores indicate that physical function, social functionality, mental health, energy/vitality and general health sub-dimensions increase. Similarly, higher scores indicate a decrease in physical role difficulty, emotional role difficulty and pain.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammet Ali AYDIN, Ph. D, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided